CLINICAL TRIAL: NCT01678378
Title: School Health Center Healthy Adolescent Relationship Program
Acronym: SHARP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12020646
Record Dates: First submitted 2012-08-30; First posted 2012-09-05 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Adolescent Relationship Abuse
Keywords: Adolescent; Intervention; Female; Male; Interpersonal Relations; School Health Services; Community-Based Participatory Research; Randomized Controlled Trial; Health Care Provider; Training Program; Harm Reduction; Prevention; Reproductive Coercion; Tech-Based Abuse; Social Environment; Sexual Partners
MeSH Terms: conditions — Harm Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SHARP Intervention (Experimental): School health centers randomized to the SHARP Intervention will be trained to address adolescent relationship abuse with school health center clients.
  Interventions: Behavioral: SHARP Intervention
- Control (No Intervention): School health centers randomized to Control will provide standard of care.

INTERVENTIONS:
Behavioral: SHARP Intervention — Providers and staff located in high school school health centers (i.e., nurse practitioners, nurses,physicians, health educators, medical assistants) will be trained to address adolescent relationship abuse with school health center clients using knowledge, skills, and resources gained through the SHARP Intervention training. The training includes strategies to help youth recognize adolescent relationship abuse among themselves and their peers, to learn strategies to increase safety (harm reduction), and to utilize adolescent relationship abuse-related resources.
  Arms: SHARP Intervention

SUMMARY:
This community-partnered participatory study will work within high school health centers (SHCs) to test, via a 2-armed cluster randomized controlled trial, a multi-level intervention to reduce adolescent relationship abuse (ARA) among adolescents ages 14-19. The goal of this study is to examine the effectiveness of the School Health Center Healthy Adolescent Relationships Program (SHARP) intervention in SHCs on individual SHC clients, the SHC clinic environment, and the schools in which the SHCs are located. Evaluation of the intervention will involve random assignment of eight comparable SHCs in the Greater Bay Area of California that provide comprehensive health services, to either intervention or control sites. Adolescent females and males ages 14-19 seeking care at any of these SHCs (N=1200) will be assessed via audio computer-assisted survey instrument (ACASI) at baseline and 16-20 weeks follow-up to examine intervention effects on knowledge and self-efficacy regarding ARA, harm reduction and ARA-related resources as well as intentions to intervene with peers. For youth reporting recent ARA victimization, the investigators will assess for increases in ARA disclosure, resource utilization, as well as reduction in ARA victimization.

ELIGIBILITY:
Inclusion Criteria:

* age 14-19
* receiving services at one of the eight SHARP Intervention school health centers
* able to read English or Spanish

Exclusion Criteria:

* clients not of the specified age range
* clients who are intoxicated or otherwise not able to provide their own consent

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1012 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Recognition of adolescent relationship abuse | 4 months
  "Recognition of abusive behaviors" -- Between-arm adjusted mean differences on a 9-item summary scale
Intentions to positively intervene in adolescent relationship abuse among peers | 4 months
  "Intentions to intervene" -- Between-arm adjusted mean differences on a 9-item summary scale
Knowledge of violence victimization resources | 4 months
  "Knowledge of resources" -- Between arm differences of summary score of single items which assess the extent to which participants are aware of places they could go for specific support services.

SECONDARY OUTCOMES:
Disclosure of adolescent relationship abuse to school health center providers | baseline (after clinic visit)
  Between-arm adjusted differences in proportion disclosing adolescent relationship abuse (ARA) to school health providers at baseline. Comparisons restricted to subgroup of clients reporting ARA on ACASI survey at baseline.
Uptake of adolescent relationship abuse harm reduction and utilization of resources | 4 months
  Between-arm adjusted differences in proportion reporting any use of ARA resources in the 3-month period prior to the follow-up survey. Comparisons restricted to clients reporting ARA on ACASI survey at baseline.
Adolescent relationship abuse victimization | 4 months
  Between-arm adjusted differences in proportion screened positive for at least one adolescent relationship abuse (ARA) behavior, based on screening tests for reproductive coercion, intimate partner and sexual violence victimization and psychological abuse. Comparisons restricted to clients reporting ARA at baseline.
Knowledge of harm reduction strategies | 4 months
  Participants are presented with a series of harm reduction behaviors to reduce risk for ARA, and asked to what extent they are aware of these strategies and self-efficacy in enacting these behaviors based on a 7-point Likert-type scale

CONTACTS AND LOCATIONS:
Overall Officials: Sandi Goldstein, Principal Investigator — Pubic Health Institute; Elizabeth Miller, MD, PhD, Principal Investigator — University of Pittsburgh, Children's Hospital of Pittsburgh of UPMC
Locations (1):
- Public Health Institute, Oakland, California, United States

REFERENCES:
- [Result] Miller E, Goldstein S, McCauley HL, Jones KA, Dick RN, Jetton J, Silverman JG, Blackburn S, Monasterio E, James L, Tancredi DJ. A school health center intervention for abusive adolescent relationships: a cluster RCT. Pediatrics. 2015 Jan;135(1):76-85. doi: 10.1542/peds.2014-2471. Epub 2014 Dec 22. PMID 25535265
- [Result] Dick RN, McCauley HL, Jones KA, Tancredi DJ, Goldstein S, Blackburn S, Monasterio E, James L, Silverman JG, Miller E. Cyber dating abuse among teens using school-based health centers. Pediatrics. 2014 Dec;134(6):e1560-7. doi: 10.1542/peds.2014-0537. Epub 2014 Nov 17. PMID 25404724
- [Result] McCauley HL, Dick RN, Tancredi DJ, Goldstein S, Blackburn S, Silverman JG, Monasterio E, James L, Miller E. Differences by sexual minority status in relationship abuse and sexual and reproductive health among adolescent females. J Adolesc Health. 2014 Nov;55(5):652-8. doi: 10.1016/j.jadohealth.2014.04.020. Epub 2014 Jun 21. PMID 24962502
- [Derived] Hill AL, Jones KA, McCauley HL, Tancredi DJ, Silverman JG, Miller E. Reproductive Coercion and Relationship Abuse Among Adolescents and Young Women Seeking Care at School Health Centers. Obstet Gynecol. 2019 Aug;134(2):351-359. doi: 10.1097/AOG.0000000000003374. PMID 31306331
- See also: U.S. Department of Justice Final Report — https://www.ncjrs.gov/pdffiles1/nij/grants/248640.pdf